CLINICAL TRIAL: NCT04924933
Title: Evaluation of Episodic Memory and Accelerated Long-term Forgetting in Patients With Drug-resistant Focal Epilepsy
Brief Title: Evaluation of Memory and Forgetting in Patients With Epilepsy
Acronym: EPIMNESIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL21_0264; 2021-A01075-36 (Other: IDRCB)
Record Dates: First submitted 2021-05-27; First posted 2021-06-14 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-01

CONDITIONS: Epilepsy
Keywords: Temporal lobe epilepsy; Episodic memory; Accelerated long-term forgetting
MeSH Terms: conditions — Epilepsy; Epilepsy, Temporal Lobe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Epilepsy group) (Experimental): Patients with drug-resistant focal epilepsy in whom an accelerated long-term forgetting is suspected (presence of a subjective memory complaint and absence of objective deficit in memory tests conducted in the frame of a routine comprehensive neuropsychological assessment)
  Interventions: Diagnostic Test: Computerised associative memory task using abstract words and landscape photographs
- Healthy volunteers (control group) (Active Comparator): Age-matched healthy volunteers
  Interventions: Diagnostic Test: Computerised associative memory task using abstract words and landscape photographs

INTERVENTIONS:
Diagnostic Test: Computerised associative memory task using abstract words and landscape photographs — Two test sessions using the computerised associative memory task will be performed by the two groups (patients and control subjects). The first session will consist of the encoding of 56 associations between a word and a photograph and the recall of half of them (28) 30 minutes later by the mean of a matching task and a recognition task. The second session consists of the recall of the other half of the associations (28) 72 hours after the encoding phase, using the same procedure (matching task and recognition task). Performance obtained by patients and by healthy volunteers will then be compared.

SUMMARY:
Drug-resistant focal epilepsy (DRFE) is frequently associated with complications of varying severity that impair patient's quality of life. Among these complications, cognitive disturbances and especially episodic memory difficulties, play a determinant part. Episodic memory can be defined as a function that allows the mental reconstruction of a past life episode, through complex associative mechanisms that link the vivid experience to its context of occurrence, called encoding context. It is a dynamic cognitive function, which calls on a widely distributed cerebral network, mainly involving the medial temporal lobe, particularly the hippocampus. Epilepsy could have a specific impact on this crucial network, disrupting the binding mechanisms between the experienced events and their encoding context, which are essential for efficient memory. Although patients with DRFE frequently demonstrate memory impairment as assessed by standardised neuropsychological tests, it only imperfectly reflects their difficulties. As a matter of fact, despite a subjective memory complaint, about 20% have no memory impairment on these tests, resulting from a phenomenon called accelerated long-term forgetting (ALF). ALF is indeed characterised by normal performance on standardised neuropsychological tests involving retention delays of 20-30 minutes, but disabling memory complaint and abnormally marked forgetting within hours or days that follow the learning period. This phenomenon is widely described at the conceptual level, but remains difficult to measure in daily practice, at least partly due to methodological limits. Thus, the validated tools available in clinical routine are poorly adapted to the complexity and the associative dimension of memory networks. There is therefore a clinical need for a specific assessment tool that would be able to detect ALF, in order to better quantify it and to enable the appropriate care of patients suffering from DRFE. The aim of the EPIMNESIE study is to evaluate the diagnostic capacity of a behavioural associative memory task, based on the analysis of encoding and consolidation mechanisms, in order to measure ALF. In this prospective study, 40 patients with DRFE and 40 healthy subjects will be proposed to complete a new associative memory task involving a learning phase and two recall sessions which will take place at 30 minutes and 72 hours after the learning phase.

ELIGIBILITY:
Epilepsy group :

Inclusion Criteria:

* Adult (≥ 18 years old) suffering from drug-resistant focal epilepsy
* Patient who recently benefit from a comprehensive neuropsychological assessment (≤2 years)
* Patient presenting a subjective memory complaint consistent with an ALF
* Patient who obtained normal performance at memory tests during the comprehensive neuropsychological assessment
* Patient who gave its written informed consent to participate to the study
* Patient with corrected or non-corrected visual acuity allowing fluid reading on a computer screen
* Patient affiliated to the French health care system

Exclusion Criteria:

* Patient with impaired reading or understanding
* Patient suffering from a major depressive syndrome (score >15 on the French version of the Neurological Disorders Depression Inventory for Epilepsy - NDDIE)
* Patient who have undergone epilepsy surgery
* Patient who presented a seizure within the hour preceding the first test session
* Protected major
* Pregnant or breastfeeding woman

Control group

Inclusion Criteria:

* Adult (≥ 18 years old) without any neurological or psychiatric history
* Adult who gave its written informed consent to participate to the study
* Adult with corrected or non-corrected visual acuity allowing fluid reading on a computer screen
* Adult with normal scores on the Montreal Cognitive Assessment (MoCA) and the Matrix reasoning sub-test of the Fourth Edition Wechsler Adult Intelligence Scale (MoCA ≥ 27/30, Matrix reasoning >5)

Exclusion Criteria:

* Adult suffering from a depressive syndrome or a significative anxiety (score ≥ 8 in each dimension of the French version of the Hospital Anxiety and Depression Scale - HADS)
* Adult presenting a spontaneous subjective memory complaint
* Protected major
* Pregnant or breastfeeding woman

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of memory loss | 30 minutes and 72 hours
  Memory loss 72 hours after the encoding phase compared to the performance obtained at 30 minutes, based on the number of correct hits (CH - calculated on 28 items) obtained at these two moments. The memory loss will be calculated as the difference between the number of CH: CH 30 minutes - CH 72 hours.

SECONDARY OUTCOMES:
Evaluation of episodic memory | 30 minutes and 72 hours
  Number of correct hits (CH) at 30-minutes and 72-hours in the Epilepsy group compared to the Control group
Qualitative distribution of errors at 30-minutes and 72-hours recalls | 30 minutes and 72 hours
  Number of false-alarm errors (FA) involving familiar but non associated items (FNAI) and number of FA involving hybrid items (HI) during the 30-minutes and 72-hours recalls in the Epilepsy group compared to the Control group
Relationship between the extent of forgetting at 30 minutes and 72 hours and the nature of contextual associations during the acquisition phase | 30 minutes and 72 hours
  Proportion of FA regarding associations categorized as "not linked" during the encoding phase
Relevance of a simple recognition to assess episodic memory at 30 minutes and 72 hours | 30 minutes and 72 hours
  Number of correct recognitions (CR) during the 30-minutes and 72-hours recalls in the Epilepsy group compared to the Control group
Effect of antiepileptic treatment currently taken by the patient (reported through clinical data) on the extent of memory loss assessed at 72 hours | 72 hours
  Relation between the number of antiseizure drugs (molecules) currently taken by the patient and available in clinical data and the memory loss (number of correct answers at 30 minutes - number of correct answers at 72 hours)
Effect of the usual frequency of seizures reported by the patient through a dedicated agenda on the extent of memory loss assessed at 72 hours | 72 hours
  Relation between monthly seizures frequency within the 3 months preceding the inclusion and reported through a dedicated agenda and the memory loss (number of correct answers at 30 minutes - number of correct answers at 72 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Guinet, PhD student, Principal Investigator — Service de Neurologie Fonctionnelle et d'Epileptologie
Locations (1):
- Hospices Civils de Lyon Service de Neurologie Fonctionnelle et d'Epileptologie, Bron, France